CLINICAL TRIAL: NCT07283523
Title: The Use of Virtual Reality to Combat Weight-Based Implicit Bias Among Physicians in Training at Brigham and Women's Hospital: A Pilot Study
Brief Title: Virtual Reality to Combat Weight-Based Implicit Bias: BWH Pilot Study
Acronym: BWH-VR-1
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Daniel Palazuelos, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P001287
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Implicit Bias; Implicit Association Test
Keywords: Reality, Virtual; Virtual Reality, Educational; Implicit Association Test; Weight-based Implicit Bias
MeSH Terms: conditions — Bias, Implicit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Encounters VR Videos (Experimental)
  Interventions: Behavioral: 360 Video on a Virtual Reality Headset
- Control Neutral VR Video (Other)
  Interventions: Behavioral: 360-Control Video

INTERVENTIONS:
Behavioral: 360 Video on a Virtual Reality Headset — Two 360- videos watched via a VR headset where the study subject will witness a positive physician encounter with a compliant obese patient and a negative encounter with a non-compliant non-obese patient
  Arms: Clinical Encounters VR Videos
Behavioral: 360-Control Video — A neutral education video from the New England Journal of Medicine watched in a 360-theatre setting via a VR headset
  Arms: Control Neutral VR Video

SUMMARY:
The goal of this pilot implementation study is to evaluate the impact of a virtual reality (VR) intervention on implicit bias for resident physicians. The main question it aims to answer are:

Does watching VR experience of two clinical encounters reduce implicit bias association test scores? Is the VR experience an acceptable intervention tool for reducing implicit bias?

Researchers will compare weight-based VR experiences consisting of two observed clinical encounters to a neutral education VR encounter to see if our intervention significantly impacts implicit bias association scores.

Participants will be asked

1. Complete Implicit Association test for weight-based bias pre-intervention and post-intervention (immediately, at one week, and one month after the intervention) to assess their implicit bias
2. Watch either experimental clinical encounter videos or neutral education video using a VR headset
3. Participants will also complete an abbreviated IAT related to views on compliance

ELIGIBILITY:
Inclusion Criteria:

* Resident physicians associated with Brigham and Women's Hospital
* Resident physicians providing informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Implicit Association Test | From enrollment to one-month post-intervention
  Participants in both experimental and control arms will take four implicit association tests: one pre-VR to assess baseline, immediately post-VR, one-week, and one-month. Impact of VR experimental experience will be assessed for significant changes in IAT scores between the pre-VR test and the post-VR tests.

SECONDARY OUTCOMES:
Resident Impression of Virtual Reality Implicit Bias Project | One-month post-VR
  The acceptability of the use of virtual reality for implicit bias studies will be surveyed

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shared since IAT scores of residents may be considered private information that a resident physician may not want shared.

REFERENCES:
- [Background] Marini M, Waterman PD, Breedlove E, Chen JT, Testa C, Reisner SL, Pardee DJ, Mayer KH, Krieger N. The target/perpetrator brief-implicit association test (B-IAT): an implicit instrument for efficiently measuring discrimination based on race/ethnicity, sex, gender identity, sexual orientation, weight, and age. BMC Public Health. 2021 Jan 19;21(1):158. doi: 10.1186/s12889-021-10171-7. PMID 33468085
- [Background] Gonzalez-Liencres C, Zapata LE, Iruretagoyena G, Seinfeld S, Perez-Mendez L, Arroyo-Palacios J, Borland D, Slater M, Sanchez-Vives MV. Being the Victim of Intimate Partner Violence in Virtual Reality: First- Versus Third-Person Perspective. Front Psychol. 2020 May 8;11:820. doi: 10.3389/fpsyg.2020.00820. eCollection 2020. PMID 32457681
- [Background] Banakou D, Slater M. Body ownership causes illusory self-attribution of speaking and influences subsequent real speaking. Proc Natl Acad Sci U S A. 2014 Dec 9;111(49):17678-83. doi: 10.1073/pnas.1414936111. Epub 2014 Nov 24. PMID 25422444
- [Background] Salmanowitz N. The impact of virtual reality on implicit racial bias and mock legal decisions. J Law Biosci. 2018 Apr 19;5(1):174-203. doi: 10.1093/jlb/lsy005. eCollection 2018 May. PMID 29707220
- [Background] Banakou D, Kishore S, Slater M. Virtually Being Einstein Results in an Improvement in Cognitive Task Performance and a Decrease in Age Bias. Front Psychol. 2018 Jun 11;9:917. doi: 10.3389/fpsyg.2018.00917. eCollection 2018. PMID 29942270
- [Background] Peck TC, Seinfeld S, Aglioti SM, Slater M. Putting yourself in the skin of a black avatar reduces implicit racial bias. Conscious Cogn. 2013 Sep;22(3):779-87. doi: 10.1016/j.concog.2013.04.016. Epub 2013 May 28. PMID 23727712
- [Background] Bertrand P, Guegan J, Robieux L, McCall CA, Zenasni F. Learning Empathy Through Virtual Reality: Multiple Strategies for Training Empathy-Related Abilities Using Body Ownership Illusions in Embodied Virtual Reality. Front Robot AI. 2018 Mar 22;5:26. doi: 10.3389/frobt.2018.00026. eCollection 2018. PMID 33500913
- [Background] Marini M, Rubichi S, Sartori G. The role of self-involvement in shifting IAT effects. Exp Psychol. 2012;59(6):348-54. doi: 10.1027/1618-3169/a000163. PMID 22750742
- [Background] Lai CK, Marini M, Lehr SA, Cerruti C, Shin JE, Joy-Gaba JA, Ho AK, Teachman BA, Wojcik SP, Koleva SP, Frazier RS, Heiphetz L, Chen EE, Turner RN, Haidt J, Kesebir S, Hawkins CB, Schaefer HS, Rubichi S, Sartori G, Dial CM, Sriram N, Banaji MR, Nosek BA. Reducing implicit racial preferences: I. A comparative investigation of 17 interventions. J Exp Psychol Gen. 2014 Aug;143(4):1765-85. doi: 10.1037/a0036260. Epub 2014 Mar 24. PMID 24661055
- [Background] Tappolet C, Teroni, F, Ziv, AK. Shadows of the Soul: Philosophical Perspectives on Negative Emotions. 2018